CLINICAL TRIAL: NCT06706505
Title: The Effect of Mindfulness Based Art Therapy Applied to Nurses Working in a University Hospital in the Earthquake Zone on Difficulties in Emotion Regulation, Burnout and Psychological Flexibility
Brief Title: Mindfulness-Based Art Therapy for Nurses: Difficulties in Emotion Regulation, Burnout, and Psychological Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehtap Ağaç (Other)
Responsible Party: Sponsor-Investigator, Mehtap Ağaç, PhD, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GAZI-HEM-MA-01
Record Dates: First submitted 2024-11-25; First posted 2024-11-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Mental Health Wellness 1; Burnout, Professional
Keywords: art therapy; mindfulness; emotional regulation; burnout; psychological flexibility; nurses
MeSH Terms: conditions — Burnout, Professional; Emotional Regulation; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: pre-test post-test follow-up and control group experimental study
Who Masked: Outcomes Assessor
Masking Description: In randomized controlled trials, it is crucial for groups to be equal and balanced in terms of baseline characteristics. To achieve this, simple stratified randomization based on gender was used to assign nurses to the intervention and control groups. To prevent bias, both researchers and participants were blinded to group assignments until after randomization. Due to the study's nature, blinding the researcher administering the intervention and participants was not feasible. However, a pre-test was administered before randomization. A blind technique was applied with the help of an independent statistician. Participants were randomly assigned using a number generator, and a third party conducted a coin flip to determine group assignments. The data will be coded by a nursing expert to ensure the statistician remains unaware during analysis. Group codes will be revealed after data analysis to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness based art therapy (Experimental): Prior to the MBAT intervention, data collection forms were administered and randomization was performed. Following the pre-test, participants in this group will attend weekly MBAT sessions for five weeks. Post-intervention, data collection forms will be administered again. Subsequent follow-up assessments will be conducted at 3 and 6 months.
  Interventions: Behavioral: Mindfulness-based art therapy
- Therapy waiting list (No Intervention): Following the pre-test and randomization, the control group will receive follow-up assessments concurrently with the intervention group at predetermined intervals (post-intervention, 3 months, and 6 months). Upon completion of the research, the participants assigned to the control group will undergo the MBAT intervention.

INTERVENTIONS:
Behavioral: Mindfulness-based art therapy — MBAT combines art therapy and mindfulness to promote self-awareness and emotional well-being. It uses art to express thoughts and feelings, while cultivating mindfulness skills. MBAT addresses stress, anxiety, and emotional regulation. Grounded in research, it's an effective therapeutic approach.
  The mindfulness-based art therapy sessions were designed based on the literature, drawing on the researches. By integrating art therapy techniques and mindfulness practices, the sessions were developed. Expert opinions were sought from specialists in the field to ensure the content validity of the sessions, and necessary adjustments were made accordingly. The MBAT application consists of five sessions in total. Each session has a specific theme and is designed to last 90-120 minutes.
  Arms: Mindfulness based art therapy

SUMMARY:
The aim of this study is to examine the effects of mindfulness-based art therapy on the difficulties in emotional regulation, burnout, and psychological resilience levels of nurses working in the earthquake-affected region. The main questions it aims to answer are:

Does MBAT reduce the burnout levels of nurses working in the earthquake-affected region? Does MBAT reduce the emotional regulation difficulties of nurses working in the earthquake-affected region? Does MBAT increase the psychological resilience levels of nurses working in the earthquake-affected region? Researchers plan to compare the intervention group where MBAT is applied and the control group where no intervention is applied to see the effects of MBAT on nurses.

Participants :

The intervention group will receive MBAT once a week for 5 weeks. The control group will receive MBAT again after the application is completed, if they are willing.

Follow-up tests will be administered before the intervention, after it is completed, and at the 3rd and 6th months."**

DETAILED DESCRIPTION:
The nursing profession, by its very nature, involves direct interaction with individuals, creating a highly emotionally charged work environment. This necessitates nurses to understand and manage their emotional states. Emotion regulation is a process that determines when, how, and to what extent individuals experience and express their emotions. Disruptions in this process can lead to difficulties in emotion regulation, anxiety, and depression.

Nurses constantly encounter patients experiencing pain, loss, and difficulties. This can lead to emotional burnout and decreased job satisfaction among nurses. Studies have shown that difficulties in emotion regulation and low psychological flexibility contribute to burnout, depersonalization, and emotional exhaustion in nurses. On the other hand, emotion regulation training and the development of psychological flexibility skills can effectively reduce occupational stress for nurses.

Psychological flexibility is defined as the ability to cope with challenges, adapt to changing circumstances, and accept negative emotional experiences. Psychological flexibility enables individuals to better adapt to life's difficulties and improve their overall well-being. For individuals working under constant stress, such as nurses, psychological flexibility is crucial for job satisfaction, quality of life, and overall health.

Mindfulness-Based Art Therapy (MBAT) is a therapeutic approach aimed at developing emotional awareness, acceptance, mental focus, and emotional regulation skills. Combining art therapy and mindfulness techniques, MBAT can help nurses cope with emotional challenges, reduce stress levels, enhance psychological flexibility, and improve overall well-being.

Nurses' emotional regulation and psychological flexibility skills are crucial for both their own psychological well-being and the quality of care they provide. Difficulties in emotion regulation and low psychological flexibility can lead to burnout and other negative consequences. Therapeutic approaches such as Mindfulness-Based Art Therapy (MBAT) offer promising solutions to support nurses' emotional health and create more sustainable professional lives.

Study Design: This study is a randomized controlled trial with a pre-test, post-test, and follow-up design. It aims to determine the effects of mindfulness-based art therapy on nurses' difficulties in emotion regulation, burnout, and psychological flexibility.

Study Setting and Characteristics: The study will be conducted at Kahramanmaraş Sütçü İmam University Health Practices and Research Hospital, located in Kahramanmaraş, Turkey. This center provides services in various departments, including internal medicine, surgery, oncology, and psychiatry, with separate units for children and adults. Nurses at this center primarily work in inpatient units, intensive care units, operating rooms, and emergency departments. Their work schedules include both day shifts and rotating shifts.

Population and Sample: The study population consists of all nurses working at Kahramanmaraş Sütçü İmam University Health Practices and Research Hospital. Based on information obtained from the institution, the total number of nurses is 500. The sample will include nurses who meet the inclusion criteria. To determine the sample size, the G*Power program was used. The effect size was calculated based on a similar study in the literature. With an alpha level of 0.05, a power of 0.95, and an effect size of 1.109189, the total sample size was calculated to be 38 (19 in the intervention group and 19 in the control group). Considering a potential dropout rate of 10-20% as reported in previous studies, the sample size was increased by 20%, resulting in a final sample size of 23 nurses in each group.

Pilot Study: Prior to the main study, a pilot study was conducted to evaluate the feasibility of a structured mindfulness-based art therapy intervention. A group of eight volunteer nurses from the outpatient clinics and polyclinics of Kahramanmaraş Sütçü İmam University Health Practices and Research Hospital participated in this pilot intervention.

Study Implementation: The main study will be conducted at Kahramanmaraş Sütçü İmam University Health Practices and Research Hospital following the pilot study. Before the intervention, both the intervention and control groups will be administered the Participant Information Form once, and the Difficulty in Emotion Regulation Scale (Short Form), the Maslach Burnout Inventory, and the Psychological Flexibility Scale three times (pre-test: one week before the MBAT, post-test: one week after the MBAT, follow-up: 3 and 6 months after the MBAT). Following the pre-test, a 5-session MBAT will be initiated for the intervention group. Considering the effectiveness of the intervention and the characteristics of psychological counseling groups, the intervention group will be divided into subgroups. Each subgroup will receive the intervention on different days or times within the same week. After the intervention period and post-test, the MBAT will be applied to the control group.

Data Analysis: Data collected from the study will be analyzed using International Business Machines (IBM) Statistical Package for the Social Sciences (SPSS) V23. To assess normality, the Shapiro-Wilk test will be used. For normally distributed data, independent samples t-test and paired samples t-test will be employed. For non-normally distributed data, the Mann-Whitney U test and the Wilcoxon signed-rank test will be used. The relationship between variables will be examined using Spearman correlation analysis. Data will be presented as mean and standard deviation for normally distributed data and median and range for non-normally distributed data. Categorical data will be analyzed using the chi-square test and presented as frequencies and percentages.

Ethical Considerations: Ethical approval has been obtained from the Ethics Committee of Gazi University (dated 16.04.2024, number 07) and the relevant departments of Kahramanmaraş Sütçü İmam University Health Practices and Research Hospital. Permission to use the data collection tools was obtained via email from the authors who conducted the validity and reliability studies. Before the study began, participants were provided with detailed information about the study's purpose, procedures, and expected outcomes. Written informed consent was obtained from each participant in the pre-test, intervention, and control groups. The researcher conducting the study possesses the necessary qualifications and certifications to implement the intervention.

ELIGIBILITY:
Inclusion Criteria:

* To have provided active care for individuals affected by the earthquake for at least three months
* To voluntarily agree to participate in the study.

Exclusion Criteria:

* To have received or be currently receiving training or individual/group therapy in art therapy or mindfulness.
* To have a condition that would prevent them from actively participating in the sessions, comprehending the scales, and completing them.
* To fail to attend two consecutive study sessions for any reason
* To voluntarily withdraw from the study at any time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) | 7 months
  The Difficulties in Emotion Regulation Scale (DERS) was developed by Gratz and Roemer (2004) to assess emotional regulation difficulties. A shorter version was created by Bjureberg et al. (2016) and adapted into Turkish by Yiğit and Güzey Yiğit (2019). The DERS-Short Form consists of 16 items and measures five factors: acceptance, clarity, goals, strategies, and impulsivity. The acceptance subscale measures rejection of emotional responses; clarity assesses understanding emotions; goals evaluates focus on goal-directed behavior during emotional experiences; strategies measures access to emotion regulation strategies; and impulsivity evaluates control over impulses when experiencing negative emotions. Higher scores indicate greater difficulties. The scale's internal consistency (Cronbach's alpha) is 0.92, with subscale consistency ranging from 0.78 to 0.87.
Maslach Burnout Inventory (MBI) | 7 months
  The Maslach Burnout Inventory (MBI), developed by Maslach and Jackson in 1981 to measure burnout, was adapted into Turkish by Ergin in 1992. The scale consists of 22 items and utilizes a 5-point Likert scale (0: Never, 1: Very rarely, 2: Sometimes, 3: Often, 4: Always). The MBI assesses three dimensions of burnout: emotional exhaustion (items 1, 2, 3, 6, 8, 13, 14, 16, 20), depersonalization (items 5, 10, 11, 15, 22), and personal accomplishment (items 4, 7, 9, 12, 17, 18, 19, and 21). Items in the personal accomplishment subscale are reverse-coded. Higher scores on emotional exhaustion and depersonalization, and lower scores on personal accomplishment, reflect greater burnout. The Turkish version's Cronbach's alpha coefficients were 0.83 for emotional exhaustion, 0.65 for depersonalization, 0.72 for personal accomplishment, and 0.93 overall (Ergin, 1992).
The Psychological Flexibility Scale | 7 months
  The original Psychological Flexibility Scale was developed by Francis, Dawson, and Golijani Moghaddam (2016). A Turkish adaptation, consisting of 37 items, was created by Karakuş and Akbay (2020) to assess psychological flexibility in adults. The original scale contained 23 items, while the Turkish version includes 28 items across five subscales: "values and behaviors aligned with values" (items 1, 7, 9, 13, 16, 19, 21, 26, 27, 28), "being in the present moment" (8, 14, 18, 20, 22, 23, 25), "acceptance" (2, 3, 5, 6, 24), "contextual self" (4, 10, 12), and "defusion" (11, 15, 17). Items 2, 3, 5, 6, 8, 18, 20, 22, 23, 24, and 25 are reverse-scored. The scale's total score ranges from 28 to 196, with higher scores indicating greater psychological flexibility. The internal consistency reliability coefficient was 0.79.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Ağaç, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University; Sultan Ayaz Alkaya, Professor, Study Chair — Gazi University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data sharing is not desired

REFERENCES:
- [Result] Bjureberg J, Ljotsson B, Tull MT, Hedman E, Sahlin H, Lundh LG, Bjarehed J, DiLillo D, Messman-Moore T, Gumpert CH, Gratz KL. Development and Validation of a Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16. J Psychopathol Behav Assess. 2016 Jun;38(2):284-296. doi: 10.1007/s10862-015-9514-x. Epub 2015 Sep 14. PMID 27239096
- [Result] Ergin C. Doktor ve hemsirelerde tukenmislik ve Maslach tukenmislik olceginin uyarlanmasi. VII. Ulusal Psikoloji Kongresi, 22th September 1992. Ankara (Turkey).
- [Result] Maslach C, Jackson SE. Maslach Burnout Inventory--ES Form (MBI). 1981. https://doi.org/10.1037/t05190-000
- [Result] Francis AW, Dawson DL, & Golijani-Moghaddam N. The development and validation of the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT). Journal of Contextual Behavioral Science. 2016: 5(3): 134-145. https://doi.org/10.1016/j.jcbs.2016.05.003
- [Result] Karakuş S, Akbay SE. Psychological Flexibility Scale: Adaptation, Validity and Reliability Study. Mersin University Journal of the Faculty of Education. 2020: 16(1): 32-43. https://doi.org/10.17860/mersinefd.665406
- [Result] Yiğit İ, Guzey Yiğit, M. Psychometric Properties of Turkish Version of Difficulties in Emotion Regulation Scale-Brief Form (DERS-16). Current Psychology. 2019: 38: 1503-1511. https://doi.org/10.1007/s12144-017-9712-7.
- [Result] Gratz, KL, Roemer, L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment. 2004: 26: 41-54. https://doi.org/10.1023/B:JOBA.0000007455.08539.94